CLINICAL TRIAL: NCT02797795
Title: A Phase 1, Open-Label, Dose-Escalation Study Evaluating the Safety, Pharmacokinetics, and Clinical Effects of Intravenously Administered NEV801 in Subjects With Advanced Malignancies
Brief Title: A Phase 1, Open-Label, Dose-Escalation Study of NEV801, Administered to Patients With Advanced Cancers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neovia Oncology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEV801-01
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Advanced Cancer; Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- NEV801 (Experimental): Part A - Dose escalation and de-escalation for the determination of the Maximum tolerated dose. All subjects will receive NEV801 intravenously on days 1, 8, 15 and 22 during each 28-day cycle.
  Part B - Subjects will receive NEV801 at or below the highest tolerable dose from Part A.
  Interventions: Drug: NEV801

INTERVENTIONS:
Drug: NEV801 — Dose Escalation

SUMMARY:
This study is a first-in-human, multicenter, open-label, nonrandomized, dose-escalation trial to be conducted in 2 sequential parts:

* Part A (Dose Escalation) in subjects with advanced malignancies
* Part B (Dose Confirmation) in subjects with tumor type(s) to be determined by results of Part A

DETAILED DESCRIPTION:
In Part A, subjects will be treated with a 30-minute intravenous (IV) infusion of NEV801 on Days 1, 8, 15, and 22 of continuous 28-day cycles. The starting dose of NEV801 will be 20 mg/m2/dose, and the NEV801 dose will be escalated in successive cohorts of 3 subjects per dose level. In Part B, up to 3 expansion cohorts of up to 12 subjects each, defined by tumor type, will be enrolled at or below the MTD (i.e., the RP2D) of NEV801. In both parts, subjects who tolerate the drug and who do not experience progressive disease may continue to receive NEV801 at the discretion of the Investigator for up to 12 cycles. Subjects who tolerate the drug and experience clinical benefit will be eligible for further treatment in an extension protocol or through another means to be determined by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age
2. Willing and able to provide written informed consent and comply with the requirements of the study
3. Pathologically confirmed advanced malignancy for which standard therapy proven to provide clinical benefit does not exist or is no longer effective
4. Part A only: Evaluable disease, measurable either on physical examination or by imaging according to RECIST v1.1 or by informative tumor marker(s)
5. Part B only: Selected tumor type(s), as determined by results of Part A
6. Part B only: Measurable disease, using RECIST v1.1
7. ECOG performance status of 0 or 1

Exclusion Criteria:

1. Receipt of more than 5 prior regimens of cytotoxic chemotherapy (unless prior approval is granted by the Sponsor)
2. Any chemotherapy, immunomodulatory drug therapy, antineoplastic hormonal therapy, immunosuppressive therapy, corticosteroids > 20 mg/day prednisone or equivalent (unless administered to prevent contrast material reactions during radiographic procedures), or growth factor treatment (e.g., erythropoietin) within 14 days before first NEV801 dose
3. Presence of an acute or chronic toxicity of prior chemotherapy, with the exception of alopecia, that has not resolved to ≤ Grade 1, according to the NCI CTCAE v4.03
4. Radiotherapy within 28 days before the first NEV801 dose
5. Use within 7 days of the first NEV801 dose, or anticipated use, of agents that are strong inhibitors of CYP3A4, CYP1A2 and CYP2D6 enzymes (unless approved by the Sponsor) - see Section 5.6 for a list of strong CYP3A4, CYP1A2 and CYP2D6 inhibitors
6. Use of any investigational agents within 28 days of the first NEV801 dose
7. Major surgery within 28 days before the first NEV801 dose
8. Life expectancy < 12 weeks
9. Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months before the first NEV801 dose
10. History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QT corrected by the Fridericia formula (QTcF) interval to > 450 msec for males or > 470 msec for females
11. Previous malignancy other than non-squamous-cell carcinoma of skin or carcinoma in situ of the uterine cervix (unless the tumor was treated with curative intent more than 2 years before the first NEV801 dose)
12. Active bacterial, viral, or fungal infection requiring systemic therapy.
13. Known HIV infection or AIDS-related illness
14. Known active viral hepatitis
15. Presence of genetic polymorphism of UGT1A1 leading to reduced glucuronidation
16. Pregnant or lactating female
17. Women of childbearing potential, unless they agree to use 2 contraceptive methods which, in the opinion of the Investigator, are effective and adequate for that subject's circumstances while on study drug and for 3 months afterward
18. Men who partner with a woman of childbearing potential, unless they agree to use 2 effective contraceptive methods (i.e., a condom, female partner using oral, injectable, or barrier method) while on study drug and for 3 months afterward
19. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or NEV801 administration; that may interfere with the informed consent process or with compliance with the requirements of the study; or that may interfere with the interpretation of study results and, in the Investigator's opinion, would make the subject inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months

SECONDARY OUTCOMES:
Observe any antitumor effects of NEV801 | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Facility, Boston, Massachusetts
  - Research Facility, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No